CLINICAL TRIAL: NCT03072706
Title: Evaluation of X-ray, Acetabular Guides and CT in THR
Acronym: EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RK174116
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Total Hip Replacement
Keywords: hip replacement; acetabulum; anteversion; position; guide
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-centre, patient-assessor blinded, parallel-group, randomised-controlled trial
Who Masked: Outcomes Assessor
Masking Description: The patient assessor will be blinded to the patients' group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): 2D X-ray templating technology
  Interventions: Other: 2D X-ray templating technology
- Corin OPS™ (Experimental): Corin Optimised Positioning System (OPS) Dynamic Hip Analysis
  Interventions: Device: Corin OPS™

INTERVENTIONS:
Device: Corin OPS™ — The OPS Dynamic Hip Analysis is a computer software package used to generate simulations of a total joint replacement from patient imaging. The dynamic simulation is used for operative planning, including implant selection, sizing and placement; and to create custom instruments or delivery specifications referencing the patient's anatomy and bio-mechanics. The simulation can also be used for the post-operative evaluation of joint performance.
  Arms: Corin OPS™
Other: 2D X-ray templating technology — Standard care where hip replacement is planned using 2D X-ray templating software
  Other Names: Standard Care
  Arms: Standard group

SUMMARY:
Total hip replacement is one of the most successful surgical procedures of modern times, with over 80,000 performed each year in the UK. However, up to 5% of all primary hip replacements need to be revised within the first 10 years, and in many cases malposition of the acetabular (hip socket) component is implicated in the early failure.

The standard method of positioning the acetabular component is for the surgeon to be guided by a combination of the visible anatomical landmarks within the surgical field, and the wider environment of the operating theatre. The advent of 3D printing has led to the development of custom-made surgical guides which can be used during surgery, in order to assist the surgeon in the positioning of instruments and devices. These surgical guides are manufactured based on CT or MRI imaging, and are designed to clearly indicate to the surgeon the desired location and orientation of bony cuts and implant positions.

This study will test the hypothesis that an acetabular alignment guide combined with three-dimensional CT-based planning using the Corin OPS™ (Optimised Positioning System), provides more accurate component alignment following primary total hip replacement compared with the current standard treatment, with the aim of improving patient outcomes and reducing the risk of complications of total hip replacement.

DETAILED DESCRIPTION:
Total hip replacement is one of the most successful surgical procedures of modern times, with over 80,000 performed each year in the UK. The vast majority of patients experience dramatic pain relief and improvement in function for many years. Despite this, however, there remains a significant risk of complications, including dislocation, leg length discrepancy, squeaking, and premature wear and failure of the implant. It is known that such complications are more likely to occur if the acetabular component is incorrectly positioned during the surgery. Up to 5% of all primary hip replacements need to be revised within the first 10 years, and in many cases malposition of the acetabular (hip socket) component is implicated in the early failure.

The Corin OPS™ offers such a custom-made acetabular alignment guide. Prior to the patient's surgery, a CT scan of the patient's pelvis & legs is performed, and the images are used to produce a 3D computer model of the patient as they stand with a "virtual" hip replacement in place. Four additional X-rays of the pelvis and lumbar spine are also taken, with the patient adopting various predetermined "functional" positions (e.g. sitting in a chair, about to stand up). From these X-rays, the changes in the pelvic and femoral orientations can be measured for these functional positions. This data is then used to drive a simulation of the movement of the 3D computer model. The orientation of the components of the virtual hip replacement are then adjusted to optimise the biomechanical function of the joint. Once the proposed implant positions have been reviewed and approved by the surgeon, a custom-made acetabular orientation guide is 3-D printed and sterilised. During the surgery, this guide is fitted into the patient's acetabulum prior to implanting the components. Using a simple system of two sterile laser pointers, the orientation indicated by the guide can then be reproduced when the definitive acetabular component is implanted. There is no published data, however, on the accuracy of acetabular component positioning using this particular method. The standard of care in the UK for acetabular component positioning is the "freehand technique", where the surgeon is to be guided by a combination of the visible anatomical landmarks within the surgical field, and the wider environment of the operating theatre. It is important that the impact of this acetabular guide on acetabular component positioning be assessed in order to determine whether this intervention is likely to improve patient outcomes and reduce the risk of complications of total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing an elective primary unilateral total hip replacement (THR) under the care of an orthopaedic consultant at University Hospitals Coventry and Warwickshire NHS Trust
* Provision of written informed consent.
* Male or Female aged 18-70 years.
* Able and willing to comply with all study requirements.

Exclusion Criteria:

* Those patients deemed by the treating clinician as unsuitable for an uncemented primary acetabular implant for reasons such as

  1. Low demand patient
  2. Osteoporosis
  3. Significant acetabular bone loss
* Patients with significant orthopaedic deformities (eg fused knee, hip or ankle).
* Unable to undergo planning imaging (unable to stand or sit for X-rays, or to lie in a CT scanner).
* Patients currently receiving ionising radiation treatment or scans for other medical conditions.
* Previous entry in this trial (contralateral THR).
* Participation in a clinical trial of an investigational medicinal product in the last 90 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Acetabular cup anteversion angle | 6 weeks (+/- 2 weeks) post-surgery
  The difference between planned and achieved acetabular cup anteversion assessed by post-operative CT scan

SECONDARY OUTCOMES:
Hip Disability & Osteoarthritis Outcome Score (HOOS) | 6-weeks, 4- and 12-months post-surgery
  Hip Disability & Osteoarthritis Outcome Score (HOOS): a validated, patient-reported measure of hip function.
Oxford Hip Score | 6-weeks, 4- and 12-months post-surgery
  Oxford Hip Score: a validated, patient-reported measure of hip function
EQ-5D | 6-weeks, 4- and 12-months post-surgery
  EQ-5D: a standardised measure of health and economic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Richard King, MBChB, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (1):
- University Hospitals Coventry and Warwickshire, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers